CLINICAL TRIAL: NCT05234151
Title: The Newborn Early Warning Score: Een Mixed Method Onderzoek
Brief Title: The Newborn Early Warning System
Acronym: NEWS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: PXL University College (Other)
Collaborators: ZOL (Other); Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FRFO049
Record Dates: First submitted 2022-01-20; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Development Tool NEWS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NEWS — Newborn Early Warning Score

SUMMARY:
Maternity wards record daily observations such as temperature, color, urine, faeces and weight of the newborn in the baby file. There is no structure and no uniformity in recording and interpreting them and in time to notify the doctor.

Adults who become ill, have clearly observable and interpretable signs such as fever, changed heart rate, and increasing pain symptoms. Verbal communication also contributes to timely risk assessment. In newborns, this is absent and vital parameters often remain good for some time despite deterioration in health status. Changes in behavior, micturition and weight can be a sign of infection or cardiopathy. Scientific studies show that in adults and children, signs of deterioration in health status are often not recognized and not acted immediately. (Paliwoda et al., 2016)

Early Warning Score Systems are used in several hospital settings with good results. ( Jensen et al., 2017; Alam et al., 2014) However, there is no universal scale that can be used for the entire hospital population. In newborns up to 120 hours postpartum, vital parameters such as heart rate, blood pressure, and saturation are currently not part of daily monitoring unlike in other hospital populations. Physical parameters such as color, micturation, weight and behavior can be a sign of decompensation and are not included in already existing measurement tools.

The healthcare industry has been very standardizing in recent years, which increases the need for a scientifically based tools tailored to the newborn.

DETAILED DESCRIPTION:
Problem Statement. Maternity wards record daily observations such as temperature, color, urine, stool and weight of the à terme newborn in the baby file. There is no structure and no uniformity in recording and interpreting these observations, nor in when the doctor should be notified.

In adults who become ill, there are clearly observable and interpretable signs such as fever, changed heart rate, and increasing pain symptoms. Verbal communication also contributes to timely risk assessment. In newborns, this is absent and vital parameters often remain good for some time despite deterioration in health status. Changes in behavior, micturition and weight can be a sign of infection or cardiopathy. Scientific studies show that in adults and children, signs of deterioration in health status are often not recognized and not acted upon in a timely manner. (Paliwoda et al., 2016) Early Warning Score Systems are used in several hospital settings with good results. ( Jensen et al., 2017; Alam et al., 2014) However, there is no universal scale that can be used for the entire hospital population. In à terme newborns up to 120 hours postpartum, vital parameters such as heart rate, blood pressure, and saturation are currently not part of daily monitoring unlike in other hospital populations. Physical parameters such as color, micturation, weight and behavior can be a sign of decompensation and are not included in already existing measurement tools.

The healthcare industry has been very standardizing in recent years, which increases the need for a scientifically based tool tailored to the newborn.

Methodology. In a first phase, a literature review will be performed to find out which parameters and trigger scores are essential in the early detection of problems in newborns up to 120 hours postpartum. A scientifically based tool will be developed to be tested, adjusted and validated in two Limburg maternities. In a before and after measurement, 20 midwives will be interviewed via semi-structured interviews about their findings before and after the use of the tool. From the medical records, information such as parameters, warning signals and time indicators will be collected and compared.

Expected Results. The research will result in descriptive statistics on the one hand, the feedback of info from the records and on the other hand from the qualitative analysis of the feedback from the interviews.

A third intended result is to present a validated Newborn Early Warning Score that can be used in the maternity department of several hospitals. This tool can also be implemented in the midwifery training to teach students how to register, interpret and report parameters of a newborn up to 120 hours postpartum in a structured way.

ELIGIBILITY:
Inclusion Criteria:

* newborn in the maternity ward

Exclusion Criteria:

* premature baby's
* ill baby's

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A term Newborns max 120 hours old
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
NEWS | 2 years
  Newborn Early Warning Score

CONTACTS AND LOCATIONS:
Locations (1):
- PXL, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No